CLINICAL TRIAL: NCT06887010
Title: A Study to Assess the Effect of Food on ABBV-101 Pharmacokinetics When Administered as an Oral ABBV-101 Tablet Formulation in Healthy Volunteers
Brief Title: A Study to Assess How Food Affects the Movement of Oral ABBV-101 Through the Body of Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M25-721
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABBV-101: Sequence 1 (Experimental): Participants will receive ABBV-101 under fasting conditions in Period 1 and will receive ABBV-101 under non-fasting conditions in Period 2
  Interventions: Drug: ABBV-101
- ABBV-101: Sequence 2 (Experimental): Participants will receive ABBV-101 under non-fasting conditions in Period 1 and will receive ABBV-101 under fasting conditions in Period 2.
  Interventions: Drug: ABBV-101

INTERVENTIONS:
Drug: ABBV-101 — Oral: Tablet

SUMMARY:
This study will assess the effect of food (high fat) on oral ABBV-101 and how ABBV-101 moves through the body in healthy adult participants

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at the time of screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* Consumption of alcohol, grapefruit products, Seville oranges, starfruit products or quinine/tonic water within the 72-hour period prior to study treatment administration.
* Use of tobacco- or nicotine-containing products within 90 days prior to the first dose of study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 45 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment
Maximum Observed Plasma Concentration (Cmax) of ABBV-101 | Up to approximately 21 days
  Maximum observed plasma concentration (Cmax) of ABBV-101
Time to Cmax (Tmax) of ABBV-101 | Up to approximately 21 days
  Tmax of ABBV-101
Area Under the Plasma Concentration-Time Curve (AUC) of ABBV-101 | Up to approximately 21 days
  AUC of ABBV-101
Terminal Phase Elimination Half-life (t1/2) of ABBV-101 | Up to approximately 21 days
  Terminal phase elimination of half-life (t1/2) of ABBV-101

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 275921, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-721